CLINICAL TRIAL: NCT02322320
Title: Continued, Long-Term Follow-Up and Lenalidomide Maintenance Therapy for Patients on BMT CTN 0702 Protocol (BMT CTN #07LT)
Brief Title: Continued, Long-Term Follow-Up and Lenalidomide Maintenance Therapy for Patients on BMT CTN 0702 Protocol (BMT CTN 07LT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN07LT; U01HL069294-05 (NIH)
Record Dates: First submitted 2014-12-17; First posted 2014-12-23 (Estimated); Results first posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2019-09

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Lenalidomide; Maintenance Therapy; Progression; Long-term; Anti-Myeloma Agents; Hematologic Disorders
MeSH Terms: conditions — Multiple Myeloma; Disease Progression; Hematologic Diseases | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tandem Auto Transplant (Active Comparator): Initial autologous transplant followed by a second autologous transplant and lenalidomide maintenance
  Interventions: Drug: Lenalidomide
- RVD Consolidation (Active Comparator): Initial autologous transplant followed by lenalidomide, bortezomib and dexamethasone (RVD) consolidation and lenalidomide maintenance
  Interventions: Drug: Lenalidomide
- Lenalidomide Maintenance (Active Comparator): Initial autologous transplant followed by lenalidomide maintenance
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — In BMT CTN 0702, maintenance therapy with lenalidomide started at 10 mg daily for three months and increased to 15 mg daily. The duration of maintenance was three years in all treatment arms. Lenalidomide will be administered initially at the patient's last documented dose prior to discontinuation of BMT CTN 0702 lenalidomide maintenance therapy. Cycle duration is 28 days. Patients will continue lenalidomide until disease progression, or discontinuation due to toxicity, death, or withdrawal from the study.
  Other Names: Revlimid™

SUMMARY:
This study is designed to compare long-term outcomes among patients randomized on the BMT CTN 0702 protocol (NCT01109004), "A Trial of Single Autologous Transplant with or without Consolidation Therapy versus Tandem Autologous Transplant with Lenalidomide Maintenance for Patients with Multiple Myeloma". It is hypothesized that use of novel anti-myeloma agents will improve long-term progression-free survival (PFS) after high-dose melphalan followed by autologous hematopoietic cell transplantation (HCT) as compared to a second autologous transplantation.

DETAILED DESCRIPTION:
This study is designed to compare long-term outcomes among patients randomized on the BMT CTN 0702 protocol (NCT01109004). All patients who consent will be followed for death, progression, Second Primary Malignancies (SPMs), and Quality of Life (QOL). Patients who do not consent to the long-term follow-up mechanism or who have experienced progression on the BMT CTN 0702 study will be followed through the standard Center for International Blood and Marrow Transplant Research (CIBMTR) long-term follow-up mechanism. Additionally, patients who are eligible and are willing to continue with lenalidomide as maintenance therapy will be provided lenalidomide free of charge. These patients will continue to receive lenalidomide as maintenance therapy until disease progression or discontinuation due to toxicity, death, or withdrawal from the study. The endpoints assessed will include progression-free survival (PFS), overall survival (OS), event-free survival (EFS), incidence of second primary malignancies (SPM) and health quality of life (QOL).

ELIGIBILITY:
Inclusion Criteria:

Patients fulfilling the following criteria will be eligible to provide continued long-term follow-up data as part of this study:

1. Enrolled and randomized on the BMT CTN 0702 protocol.
2. Alive at the completion of BMT CTN 0702 protocol specified follow-up defined as 4 years post-randomization.
3. Patients without evidence of disease progression at the completion of BMT CTN 0702 protocol specified follow up.
4. Signed Informed Consent Form.
5. Patients with the ability to speak English or Spanish are eligible to participate in the HQL component of this trial.

Inclusion Criteria for Optional Long-term Lenalidomide Maintenance Therapy:

Patients fulfilling the following criteria will be eligible to provide continued long-term follow-up data AND receive long-term lenalidomide maintenance therapy as part of this study:

1. Enrolled and randomized to BMT CTN 0702.
2. Completion of 3 years of maintenance therapy on BMT CTN 0702.
3. Registered in the mandatory Revlimid REMS® program (formerly the RevAssist® for Study Participants (RASP) program), and be willing and able to comply with the requirements of the Revlimid REMS® program, including counseling, pregnancy testing, and phone surveys.
4. Signed informed consent form.
5. Patients with the ability to speak English or Spanish are eligible to participate in the HQL component of this trial.

Exclusion Criteria:

Patients who meet any of the following criteria will be ineligible to receive long-term lenalidomide maintenance therapy as part of this study:

1. Patients who have evidence of disease progression prior to enrollment.
2. Patients who were discontinued from BMT CTN 0702 lenalidomide maintenance therapy, for any reason, prior to the completion of the 3 years of 0702 maintenance.
3. Female patients who are pregnant (positive - Beta Human Chorionic Gonadotropin) or breastfeeding.
4. Females of childbearing potential (FCBP) or men who have sexual contact with FCBP unwilling to use contraceptive techniques during the length of lenalidomide maintenance therapy.
5. Patients who experienced thromboembolic events while on full anticoagulation during prior therapy with lenalidomide.
6. Patients unwilling to take Deep Vein Thrombosis (DVT) prophylaxis.
7. Patients who developed a second primary malignancy, excluding non-melanoma skin cancers after initiation of lenalidomide maintenance therapy on BMT CTN 0702.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, Study Director — Center for International Blood and Marrow Transplant Research
Locations (42):
- United States (42):
  - Arizona Cancer Center, Tucson, Arizona
  - City of Hope National Medical Center, Duarte, California
  - University of California, San Diego Medical Center, La Jolla, California
  - Stanford Hospital and Clinics, Stanford, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Florida College of Medicine, Gainesville, Florida
  - University of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - BMT Group of Georgia (Northside Hospital), Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Hospital, Kansas City, Kansas
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - DFCI, Brigham and Womens Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute/BMT, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, Barnes Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Center, Buffalo, New York
  - North Shore University Hospital, Lake Success, New York
  - Mount Sinai Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of North Carolina Hospital at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Jewish Hospital BMT Program, Cincinnati, Ohio
  - University Hospitals of Cleveland/Case Western, Cleveland, Ohio
  - Ohio State/Arthur G. James Cancer Hospital, Columbus, Ohio
  - University of Oklahoma Medical Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Penn State College of Medicine, The Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Blood & Marrow Transplant Program, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas/MD Anderson CRC, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - West Virginia University Hospital, Morgantown, West Virginia
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript and supporting information submitted to NIH BioLINCC (including data dictionaries, case report forms, data submission documentation, documentation for outcomes dataset, etc where indicated).
Supporting Information: Study Protocol, ICF
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- See also: National Marrow Donor Program — http://bethematch.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tandem Auto Transplant | RVD Consolidation | Lenalidomide Maintenance
Started | 98 | 86 | 89
Completed | 98 | 86 | 89
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tandem Auto Transplant | RVD Consolidation | Lenalidomide Maintenance | Total
Number analyzed (Participants) | 98 | 86 | 89 | 273
Age, Continuous [Median (Full Range); unit: years] | 55 [28 to 70] | 56 [28 to 69] | 57 [31 to 66] | 56 [28 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 31 | 34 | 105
  Male | 58 | 55 | 55 | 168
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 5 | 2 | 18
  Not Hispanic or Latino | 81 | 77 | 84 | 242
  Unknown or Not Reported | 6 | 4 | 3 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 5 | 4 | 11
  Black or African American | 22 | 10 | 16 | 48
  White | 68 | 69 | 68 | 205
  Multiracial | 2 | 0 | 1 | 3
  Other | 1 | 0 | 0 | 1
  Unknown or Not Reported | 3 | 2 | 0 | 5
Karnofsky Performance Score (KPS) [Count of Participants; unit: Participants] — KPS describes patient-perceived global quality of life and functioning on a scale of 0-100.
  100: No evidence of disease; 90: Normal activity. Minor signs or symptoms of disease; 80: Normal activity with effort. Some signs or symptoms of disease; 70: Cares for self. Unable to continue normal activity; 60: Needs occasional assistance, but cares for most personal needs; 50: Needs considerable assistance and medical care; 40: Disabled. Needs special care and assistance; 30: Severely disabled. Hospital admission indicated; 20: Very sick. Active supportive therapy needed; 10: Moribund; 0: Dead
  Participants
    90-100 | 78 | 60 | 63 | 201
    70-80 | 20 | 26 | 26 | 72
Diseae Risk at BMT CTN 0702 Enrollment [Count of Participants; unit: Participants] — Participants on this study will be stratified for the purposes of statistical analysis into high-risk and standard risk-groups. High-risk multiple myeloma is defined by the presence of high beta-2 microglobulin (> 5.5mg/L) or the presence of cytogenetic abnormalities including t(4;14), t(14;20), t(14;16), deletion (17p) detected by FISH or standard cytogenetics, deletion 13 detected by standard cytogenetics only or aneuploidy. Participants without cytogenetic analysis available and beta-2 microglobulin ≤ 5.5mg/L or with deletion 13 detected by FISH will be classified as standard-risk disease.
  Participants
    Standard | 73 | 65 | 72 | 210
    High | 25 | 21 | 17 | 63

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression-free Survival (PFS)
Description: This analysis includes all randomized subjects from the BMT CTN 0702 protocol classified according to their randomized treatment assignment (intention-to-treat). Progression-free survival is defined as survival without disease progression or initiation of non-protocol anti-myeloma therapy. To account for loss to follow-up, the Kaplan-Meier estimator was used to estimate progression-free survival during the 5 year post-randomization follow-up period.
Time Frame: 5 years post-randomization in BMT CTN 0702
Population: All 754 randomized BMT CTN 0702 participants are included in this analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tandem Auto Transplant | RVD Consolidation | Lenalidomide Maintenance
Number analyzed (Participants) | 247 | 254 | 257
percentage of participants | 47.7 [41.1 to 53.8] | 44.1 [38.0 to 50.3] | 45.0 [38.8 to 51.2]
Statistical Analysis 1: Comparison: Tandem Auto Transplant vs RVD Consolidation; The null hypothesis is that the percentages of participants with PFS at 5 years post-randomization in BMT CTN 0702 are equal for those assigned to Tandem auto transplant and RVD consolidation therapy; Test type: Superiority; p = 0.60, Log Rank — The primary analysis involved pairwise comparisons of PFS between the three treatment arms. To control the familywise type I error rate at 0.05, two-sided testing was performed at a Bonferroni-adjusted significance level of 0.0167 = 0.05 / 3; The log rank test was stratified on risk status at BMT CTN 0702 enrollment (high risk vs. standard risk)
Statistical Analysis 2: Comparison: Tandem Auto Transplant vs Lenalidomide Maintenance; The null hypothesis is that the percentages of participants with PFS at 5 years post-randomization in BMT CTN 0702 are equal for those assigned to Tandem auto transplant and Lenalidomide maintenance therapy; Test type: Superiority; p = 0.35, Log Rank — [p-value comment as in outcome 1, analysis 1]; The log rank test was stratified on risk status at BMT CTN 0702 enrollment (high risk vs. standard risk)
Statistical Analysis 3: Comparison: RVD Consolidation vs Lenalidomide Maintenance; The null hypothesis is that the percentages of participants with PFS at 5 years post-randomization in BMT CTN 0702 are equal for those assigned to RVD consolidation and Lenalidomide maintenance therapy; Test type: Superiority; p = 0.68, Log Rank — [p-value comment as in outcome 1, analysis 1]; The log rank test was stratified on risk status at BMT CTN 0702 enrollment (high risk vs. standard risk)

2. Secondary Outcome: Percentage of Participants With Overall Survival (OS)
Description: This analysis includes all randomized subjects from the BMT CTN 0702 protocol classified according to their randomized treatment assignment (intention-to-treat). Overall survival is defined as survival of death from any cause. To account for loss to follow-up, the Kaplan-Meier estimator was used to estimate overall survival during the 5 year post-randomization follow-up period.
Time Frame: 5 years post-randomization in BMT CTN 0702
Population: All 754 randomized BMT CTN 0702 participants are included in this analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tandem Auto Transplant | RVD Consolidation | Lenalidomide Maintenance
Number analyzed (Participants) | 247 | 254 | 257
percentage of participants | 74.7 [69.1 to 80.0] | 75.4 [70.0 to 80.6] | 76.4 [71.0 to 81.5]
Statistical Analysis 1: Comparison: Tandem Auto Transplant vs RVD Consolidation; The null hypothesis is that the percentages of participants with OS at 5 years post-randomization in BMT CTN 0702 are equal for those assigned to Tandem auto transplant and RVD consolidation therapy; Test type: Superiority; p = 0.57, Log Rank — The analysis involved pairwise comparisons of OS between the three treatment arms. To control the familywise type I error rate at 0.05, two-sided testing was performed at a Bonferroni-adjusted significance level of 0.0167 = 0.05 / 3; The log rank test was stratified on risk status at BMT CTN 0702 enrollment (high risk vs. standard risk)
Statistical Analysis 2: Comparison: Tandem Auto Transplant vs Lenalidomide Maintenance; The null hypothesis is that the percentages of participants with OS at 5 years post-randomization in BMT CTN 0702 are equal for those assigned to Tandem auto transplant and Lenalidomide maintenance therapy; Test type: Superiority; p = 0.38, Log Rank — [p-value comment as in outcome 2, analysis 1]; The log rank test was stratified on risk status at BMT CTN 0702 enrollment (high risk vs. standard risk)
Statistical Analysis 3: Comparison: RVD Consolidation vs Lenalidomide Maintenance; The null hypothesis is that the percentages of participants with OS at 5 years post-randomization in BMT CTN 0702 are equal for those assigned to RVD consolidation and Lenalidomide maintenance therapy; Test type: Superiority; p = 0.77, Log Rank — [p-value comment as in outcome 2, analysis 1]; The log rank test was stratified on risk status at BMT CTN 0702 enrollment (high risk vs. standard risk)

3. Secondary Outcome: Percentage of Participants With Event-free Survival (EFS)
Description: This analysis includes all randomized subjects from the BMT CTN 0702 protocol classified according to their randomized treatment assignment (intention-to-treat). Event-free survival is defined as survival without disease progression, second primary malignancy, and death. To account for loss to follow-up, the Kaplan-Meier estimator was used to estimate event-free survival during the 5 year post-randomization follow-up period.
Time Frame: 5 years post-randomization in BMT CTN 0702
Population: All 754 randomized BMT CTN 0702 participants are included in this analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tandem Auto Transplant | RVD Consolidation | Lenalidomide Maintenance
Number analyzed (Participants) | 247 | 254 | 257
percentage of participants | 44.2 [38.0 to 50.5] | 42.1 [36.1 to 48.3] | 42.4 [36.4 to 48.6]
Statistical Analysis 1: Comparison: Tandem Auto Transplant vs RVD Consolidation; The null hypothesis is that the percentages of participants with EFS at 5 years post-randomization in BMT CTN 0702 are equal for those assigned to Tandem auto transplant and RVD consolidation therapy; Test type: Superiority; p = 0.67, Log Rank — The analysis involved pairwise comparisons of EFS between the three treatment arms. To control the familywise type I error rate at 0.05, two-sided testing was performed at a Bonferroni-adjusted significance level of 0.0167 = 0.05 / 3; The log rank test was stratified on risk status at BMT CTN 0702 enrollment (high risk vs. standard risk)
Statistical Analysis 2: Comparison: Tandem Auto Transplant vs Lenalidomide Maintenance; The null hypothesis is that the percentages of participants with EFS at 5 years post-randomization in BMT CTN 0702 are equal for those assigned to Tandem auto transplant and Lenalidomide maintenance therapy; Test type: Superiority; p = 0.20, Log Rank — [p-value comment as in outcome 3, analysis 1]; The log rank test was stratified on risk status at BMT CTN 0702 enrollment (high risk vs. standard risk)
Statistical Analysis 3: Comparison: RVD Consolidation vs Lenalidomide Maintenance; The null hypothesis is that the percentages of participants with EFS at 5 years post-randomization in BMT CTN 0702 are equal for those assigned to RVD consolidation and Lenalidomide maintenance therapy; Test type: Superiority; p = 0.40, Log Rank — [p-value comment as in outcome 3, analysis 1]; The log rank test was stratified on risk status at BMT CTN 0702 enrollment (high risk vs. standard risk)

4. Secondary Outcome: Percentage of Participants With Secondary Primary Malignancies (SPM)
Description: This analysis includes all randomized subjects from the BMT CTN 0702 protocol classified according to their randomized treatment assignment (intention-to-treat). SPM is defined as development of any second malignancy, excluding non-melanoma skin cancers. To account for loss to follow-up, the Aalen-Johansen estimator was used to estimate the cumulative incidence of SPM during the 5 year post-randomization follow-up period.
  The development of any SPMs excludes non-melanoma skin cancers. Death without SPMs will be considered a competing risk for this event. The cumulative incidence of SPMs will be compared between treatment arms.
Time Frame: 5 years post-randomization in BMT CTN 0702
Population: All 754 randomized BMT CTN 0702 participants are included in this analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tandem Auto Transplant | RVD Consolidation | Lenalidomide Maintenance
Number analyzed (Participants) | 247 | 254 | 257
percentage of participants | 10.8 [7.2 to 15.1] | 7.9 [4.9 to 11.6] | 7.2 [4.3 to 10.8]
Statistical Analysis 1: Comparison: Tandem Auto Transplant vs RVD Consolidation; The null hypothesis is that the percentages of participants with SPM at 5 years post-randomization in BMT CTN 0702 are equal for those assigned to Tandem auto transplant and RVD consolidation therapy; Test type: Superiority; p = 0.43, Gray's test — The analysis involved pairwise comparisons of SPM between the three treatment arms. To control the familywise type I error rate at 0.05, two-sided testing was performed at a Bonferroni-adjusted significance level of 0.0167 = 0.05 / 3; Gray's test was stratified on risk status at BMT CTN 0702 enrollment (high risk vs. standard risk)
Statistical Analysis 2: Comparison: Tandem Auto Transplant vs Lenalidomide Maintenance; The null hypothesis is that the percentages of participants with SPM at 5 years post-randomization in BMT CTN 0702 are equal for those assigned to Tandem auto transplant and Lenalidomide maintenance therapy; Test type: Superiority; p = 0.70, Gray's test — [p-value comment as in outcome 4, analysis 1]; Gray's test was stratified on risk status at BMT CTN 0702 enrollment (high risk vs. standard risk)
Statistical Analysis 3: Comparison: RVD Consolidation vs Lenalidomide Maintenance; The null hypothesis is that the percentages of participants with SPM at 5 years post-randomization in BMT CTN 0702 are equal for those assigned to RVD consolidation and Lenalidomide maintenance therapy; Test type: Superiority; p = 0.70, Gray's test — [p-value comment as in outcome 4, analysis 1]; Gray's test was stratified on risk status at BMT CTN 0702 enrollment (high risk vs. standard risk)

5. Secondary Outcome: Percentage of Participants With Disease Progression
Description: This analysis includes all randomized subjects from BMT CTN 0702, classified by their treatment assignment (intention-to-treat). Disease progression is defined as progression of multiple myeloma, including one or more of the following:
  * Reappearance of serum monoclonal paraprotein at a level >= 0.5 g/dL
  * 24-hour urine protein electrophoresis of at least 200mg paraprotein/24 hours
  * Abnormal free light chain levels of >10 mg/dl, only in patients without measurable paraprotein in serum and urine
  * At least 10% plasma cells in a bone marrow aspirate or trephine biopsy
  * Definite increase in the size of existing bone lesions or soft tissue plasmacytomas
  * Development of new bone lesions or soft tissue plasmacytomas
  * Development of hypercalcemia (corrected serum Ca >11.5 mg/dL or >2.8 mmol/L) not attributable to other causes
  To account for loss to follow-up, the Aalen-Johansen estimator was used to estimate the cumulative incidence of progression during the follow-up period.
Time Frame: 5 years post-randomization in BMT CTN 0702
Population: All 754 randomized BMT CTN 0702 participants are included in this analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tandem Auto Transplant | RVD Consolidation | Lenalidomide Maintenance
Number analyzed (Participants) | 247 | 254 | 257
percentage of participants | 48.8 [42.5 to 55.2] | 54.3 [48.1 to 60.4] | 54.2 [48.0 to 60.4]

ADVERSE EVENTS:
Time Frame: 22 months post-enrollment to BMT CTN 07LT
Arm/Group | Tandem Auto Transplant | RVD Consolidation | Lenalidomide Maintenance
All-Cause Mortality (participants affected / at risk) | 4/98 | 4/86 | 2/89
Serious Adverse Events (participants affected / at risk) | 6/98 | 10/86 | 6/89
Other Adverse Events (participants affected / at risk) | 0/98 | 0/86 | 0/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tandem Auto Transplant (N=98) | RVD Consolidation (N=86) | Lenalidomide Maintenance (N=89)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
B precursor type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
B-cell type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-04-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT02322320/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT02322320/SAP_001.pdf